CLINICAL TRIAL: NCT00657787
Title: Development of a Post-Traumatic Stress Disorder (PTSD) Population Registry for Veterans
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); Carelon Research (Other); Boston University (Other)
Responsible Party: Sponsor
Other Study IDs: PT075235
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Posttraumatic Stress Disorder; Veterans; Health Services
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PTSD: Combat-exposed men and women with PTSD deployed to OIF/OEF.
- High Utilizers: A comparison group of combat veterans who are high utilizers of VA medical care, but who have not received a diagnosis of PTSD
- Not OIF/OEF: A second comparison group will consist of veterans with similar service record and demographic backgrounds, who were not deployed to the OIF/OEF war zones

SUMMARY:
The overall objective of this project is to develop the first longitudinal registry of combat-exposed men and women with PTSD. This registry will provide essential data on the natural history, including progression and remission, and outcomes associated with PTSD in military service men and women who have utilized the Department of Veterans Affairs (VA) health care system. Additional goals of this project are to determine risk factors for PTSD among combat-exposed service men and women (by incorporating a combat-exposed non-PTSD group of veterans into analyses), and to assess the joint effects of combat exposure and PTSD on a broad range of outcome measures (by incorporating a non-combat-exposed group of veterans into analyses). Thus, the registry will allow an evaluation of current theoretical models of symptom development and progression in a large sample of service men and women who utilize the VA medical system.

In addition to the PTSD registry, we will collect information on two comparison groups of OIF/OEF-era veterans to conduct nested case control studies within the general VA health care utilization database. First, a comparison group of combat veterans who are high utilizers of VA medical care, but who have not received a diagnosis of PTSD will be identified. This group will be used in analyses to identify risk factors for PTSD. Additionally, the rate of PTSD symptoms will be evaluated in this comparison group to estimate the prevalence of missed PTSD diagnoses among combat veterans with high rates of service utilization, and the resulting impact on utilization and outcomes. A second comparison group will consist of veterans with similar service record and demographic backgrounds, who were not deployed to the OIF/OEF war zones. Thus, the proposed project will create a PTSD registry from the VA database to assess the natural history and progression of PTSD in combat veterans from OIF/OEF and also to conduct case-control studies nested within the VA database. The case-control comparisons will be used to evaluate key hypotheses related to the specific aims of the overall project.

DETAILED DESCRIPTION:
This project will be designed to address a range of research questions within the registry itself, as well as in the comparisons with non-registry groups. Specific aims of this project can be divided into the following major research areas.

1. Epidemiology of PTSD Aim 1. To evaluate the natural history of PTSD, including progression and remission of symptoms over time, and the long-term psychosocial, medical and quality of life outcomes associated with the disorder Aim 2. To identify predictors of recovery or remission from PTSD, including treatment utilization, psychiatric and medical comorbidities, and sociodemographic factors Aim 3. To identify clinical characteristics, risk factors and comorbidities of PTSD, including disparities by gender, race/ethnicity, social support, and socioeconomic status, by comparing PTSD patients to a "control" group of veterans without PTSD
2. PTSD Treatment and Outcomes Aim 4. To identify current treatment approaches and outcomes of treatment through time, particularly among service members who are often excluded from clinical trials due to comorbidities and therefore remain unexamined and possibly under-treated Aim 5. To estimate the joint effects of combat exposure and PTSD on long-term psychosocial well-being and quality of life measures, by comparing PTSD patients to a "control" group of veterans who were not deployed to combat/war zones during the same time period
3. Health Services Research Aim 6. To establish the prevalence of PTSD in a comparison group of service men and women who had not received the PTSD diagnosis in their patient record but are high utilizers of the VA medical system, and to identify risk factors for missed PTSD diagnoses Aim 7. To provide data that are immediately useful for determining future health services policy, costs, and needs for upcoming research, manpower and training, by assessing current referral and utilization patterns. Both direct and indirect (e.g., productivity loss, pharmacological burden) costs of treatment will be assessed Aim 8. To develop a large database of servicemen and women with PTSD and network of treatment sites that are potentially available for further observational and interventional studies, as well as concurrent ancillary studies, such as qualitative studies on caregiver/family burden.

The proposed project will be conducted in three phases over three years using both existing data from the VA medical record database and prospective data to be collected by a structured interview in the third phase of the study, as well as periodic data transfers from the medical records. During the first phase (months 1-9), the data de-identification procedures for the study will be pre-tested (months 1-2), the data will be prepared for abstraction (months 2-4), and the study protocol and research interview will be reviewed and finalized (months 6-9). During Phase II (months 4-12), the preliminary PTSD database will be created by data transfer (month 4), query reports/resolutions (month 5). Also during this phase, analyses of existing data extracted from the VA medical record system will be conducted (months 10-12) and target cohorts for follow-up assessment will be identified. Phase III (months 12-36) will include subject recruitment for the PTSD registry and two comparison groups, and the structured telephone interviews will be conducted in all three groups (months 12-24). Data collected in the telephone interview will be coded, de-identified and merged with the overall study database. Analyses will be conducted during this phase (months 24-36) related to the Specific Aims of the study. The PTSD registry database will be updated as new VA electronic medical records for registry participants appear during the course of this project, thereby capturing the trajectory of PTSD patients.

Participants and Sampling Strategy The source of participants will be the VA in/outpatient electronic medical records of all new utilizers of the VA medical system from FY 2002 through 2007. According to data from the DOD Defense Manpower Data Center (DMDC) received by the VA Environmental Epidemiology Service (EES) on April 17, 2007, from FY 2002 through February 2007, there had been a total of 717,196 unique OIF/OEF veterans (excluding 3,303 who died in theater) who had been separated from active duty following deployment, and were therefore eligible for VA benefits. Of these, 252,095 (35%) had obtained VA health care by March 2007. More recent healthcare data through September 2007 indicate that 263,909 individuals have accessed VA health care. The VA health administrative database rigorously records all in-patient and out-patient visits, and includes basic information regarding each visit, such as the patient name, SSN, DOB, gender, and ICD-9 diagnostic codes to describe the purpose of the visit (EES database).

The overarching objective of this project-the creation of a PTSD registry-will be accomplished by identifying male and female OIF/OEF veterans from the entire VA medical records database of new utilizers with a diagnosis of PTSD (as defined by ICD-9 code 309.81) in the electronic medical record. We will sample from the VA database to recruit participants for a structured telephone interview to obtain details on exposures and outcomes of interest that are not captured in the existing database. A sample of 800 PTSD patients with OIF/OEF war zone experience, 400 patients without the PTSD diagnosis but with OIF/OEF experience and high utilization of VA services, and 400 individuals matched by age, gender, race/ethnicity, and year of entry into the VA EES database, who were not sent to the war zones of OIF/OEF will be recruited to participate in the telephone interview. To be representative of all veterans from the OIF/OEF era, the sampling will be stratified by year of entry into the VA database.

Creation of the PTSD Registry Database Patient registries, as defined by the AHRQ and World Health Organization, are organized systems containing information about individual persons,42 and the patient registry database is defined as a file (or files) derived from the registry. A patient-based database is necessary to allow direct access to information on diagnoses of interest and treatment outcomes, as well as to longitudinally track follow-up visits, progress, and treatment courses.

In contrast to these criteria, the current database of utilizers of the VA healthcare system is structured by chronological in-patient and out-patient visits, rather than unique patient identifiers or diagnoses. Thus, with the existing database, there is no readily accessible way to identify unique patients with PTSD or to assess their longitudinal outcomes and utilization of VA healthcare. Therefore, a fundamental objective of this proposal is to establish a registry of patients with PTSD from the existing VA utilization database. Electronic medical records such as those in the VA database are increasingly important sources of data, but data must be extracted, transformed into registry format, and loaded into the registry, where they will reside in the registry database, together with registry-specific data that is imported from other sources. The other sources of data for the PTSD registry will be the OIF/OEF veteran roster (particularly for military specific data, e.g., branch, rank, deployment dates, etc.) and, in Phase III, the proposed telephone interview.

During Phase I of this project, a cumulative roster of unique OIF/OEF veterans who have been separated from active duty following deployment and who have become eligible for VA healthcare will be matched with VA inpatient (PTF) and outpatient (OPC) databases for fiscal year (FY) 2004 through FY 2007. For identification of a potential PTSD patient, any veteran patient with a diagnosis of ICD-9 CM, 308.81 will be selected. The PTSD registry will encompass utilizers of the VA medical system. Each unique patient with a visit record indicating a PTSD diagnosis will be included. The registry creation will involve a multi-step process, including steps to identify all PTSD diagnoses, to identify unique patients within the PTSD diagnoses, and to identify each additional visit made by each PTSD patient. For identification of OIF/OEF veteran non-PTSD patients who are high VA healthcare users (sample #2), we will review in/outpatient records of OIF/OEF veteran patients and identify those who have been hospitalized or treated as outpatients more than 11 times during the post deployment period. A similar step will be taken to identify a non-combat comparison group of patients (sample #3). All veteran patients for three groups will be stratified by year of first entry to VA healthcare data bases (FY 2004-2007) and equal number of veteran patients will be randomly selected for each fiscal year for sample #1 and sample #2. For sample #3, additional matching variables such as age, gender, and ethnicity/race will be used in addition to the year of entry to VA healthcare databases. Ultimately, during Phase II, all existing VA medical utilization data and OIF/OEF veterans' roster data for each veteran patient will be merged and de-identified to ensure privacy and confidentiality.

During Phase III, data obtained from a telephone interview will be merged with the existing data in the PTSD registry database. The PTSD registry will continue to be updated at 6-month intervals during the course of this project as new or updated electronic medical records are entered into the VA in/outpatient healthcare database for registry participants.

ELIGIBILITY:
Inclusion Criteria:

* Veteran

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: US Military Veterans
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2008-09; Primary Completion 2017-01 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
PTSD Diagnosis | over the course of the study
  PTSD diagnosis based on SCID-5 semi-structured interview

SECONDARY OUTCOMES:
Life Events Checklist | Past and current
  checklist of potentially traumatic experiences
Prime-MD Patient Health Questionnaire | Past and Current
  measures DSM-5 depression, GAD, Panic Disorder
Alcohol Use Disorder Identification Test (AUDIT) | past and current
  Alcohol Use Disorder screener
Defense and Veterans Brain Injury Center TBI questionnaire, modified for brief administration | Past
  screens for history of traumatic brain injury
Deployment Risk and Resilience Inventory (DRRI) Section L (Post-deployment support) | Current
  post deployment social support
Veterans RAND 12 Item Health Survey (VR-12) | Current
  a patient-reported global health measure that is used to assess a patient's overall perspective of their quality of life
Sleep Problem Scale | Current
  Sleep Quality
Treatment and Service Utilization - study specific questions | Current
  These questions focus on the extent to which participants are enrolled in and use VA and non-VA healthcare services
Inventory of Psychosocial Functioning (IPF) | Current
  self report measure of functioning across social, occupational, and other domains

CONTACTS AND LOCATIONS:
Overall Officials: Terence M Keane, PhD, Principal Investigator — BUSM; VA Boston Healthcare System
Locations (1):
- VA Boston Healthcare System (Jamaica Plain Campus), Boston, Massachusetts, United States